CLINICAL TRIAL: NCT03233399
Title: Modulating Movement Intention Via Cortical Stimulation in Healthy Subjects and Patients With Psychogenic Movement Disorders and Non-epileptic Seizures
Brief Title: Modulating Movement Intention Via Cortical Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-01859
Record Dates: First submitted 2017-07-24; First posted 2017-07-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Seizures; Seizure Disorder; Psychogenic Movement Disorder
Keywords: Electroencephalography; Magnetoencephalography; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Seizures; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Healthy Patients (Active Comparator): All healthy volunteers will complete the healthy volunteer form, MRI safety screening form, and the Montreal Cognitive Assessment (MOCA).
  Interventions: Device: Sham TMS3 stimulation; Device: rTMS of left or right angular gyrus (AG) or frontal cortex (FC); Device: Anodal tDCS of left or right AG or FC
- PMD/PNES patients (Active Comparator): PMD and PNES subjects will be referred by the treating
  Interventions: Device: Sham TMS3 stimulation; Device: rTMS of left or right angular gyrus (AG) or frontal cortex (FC); Device: Anodal tDCS of left or right AG or FC

INTERVENTIONS:
Device: Sham TMS3 stimulation — half of the subjects will receive sham stimulation first
Device: rTMS of left or right angular gyrus (AG) or frontal cortex (FC) — Half of the subjects will receive active stimulation first; A subject may receive either TMS or tDCS stimulation, but not both, over the course of the sub-study.
  Other Names: 45 Minutes
Device: Anodal tDCS of left or right AG or FC — Half of the subjects will receive active stimulation first; A subject may receive either TMS or tDCS stimulation, but not both, over the course of the sub-study.
  Other Names: 30 Minutes

SUMMARY:
The purpose of this protocol is to learn about movement intention and volition. To improve such knowledge, investigators will conduct sub-studies using multiple non-invasive methodologies. These results could provide preliminary data for subsequent studies evaluating local and global efficacy of plasticity-inducing treatments for PMD symptoms.

DETAILED DESCRIPTION:
This study will:

* Explore effects of TMS and tDCS on movement intention.
* Discern the neural activity underlying modulation of movement intention with neuroimaging recording.
* Identify brain stimulation's effect in patients with psychogenic tremor and non-epileptic seizures.
* Technical development of new experimental paradigms and data analysis methods.
* Data collection for hypotheses development.

ELIGIBILITY:
Inclusion Criteria:

(Healthy Controls)

* Fluent in English

(Patients with PMD or PNES):

* Diagnosis of PMD/PNES confirmed by a neurologist with expertise in movement disorders.
* Per the treating neurologist, subject is unlikely to require treatment and/or dosage changes for 3-6 months following screening

Exclusion Criteria:

* Any history of a significant neurological disorder, which may interfere with the interpretation of study data, as determined by the PI
* Chronic or progressive medical condition
* Any history of traumatic brain injury or significant head trauma
* Currently meets criteria for substance abuse or dependence
* History of any psychotic disorder or other psychiatric condition which may interfere with data interpretation
* Pregnancy
* Metal or devices in the head, including neurostimulators or metal foreign bodies
* Any other implanted metal device, including pacemaker, spinal cord stimulator, VNS.
* Any other ferromagnetic substance in the body that may increase study risk (including dental prosthetics, etc.).
* Taking tricyclic antidepressant or antiepileptic medications or CNS active drugs under "strong potential hazard" list in Rossi et al., 2009
* Current diagnosis of any inflammatory or autoimmune disorder within last 6 months

PMD and PNES Patients

* Any history of traumatic brain injury or significant head trauma
* Diagnosis of organic seizure disorder, including febrile seizures and tonic-clonic seizures;
* Neurological disorder other than PMD and PNES including stroke, fainting spells or syncope of unknown cause(s);
* Major or unstable medical illness, especially any current diagnosis of inflammatory or autoimmune disorders within last 6 months
* Metal or devices in the head, including neurostimulators or metal foreign bodies
* Taking tricyclic antidepressant medications or CNS active drugs under "strong potential hazard" list in Rossi et al., 2009;
* Diagnosis of dementia, or Montreal Cognitive Assessment (MoCA) ≤24;
* Recurrent visual hallucinations, within the past 6 months;
* History of significant uncontrollable movements of the head;
* Any clinically significant abnormality on vital signs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Changes in signal intensity measured using of tDCS | 30 Minutes
  as a result of altering cerebral perfusion in response to neurophysiologic stimulation
Changes in signal intensity measured during EEG recording | 3 Hours
  as a result of altering cerebral perfusion in response to neurophysiologic stimulation
Changes in signal intensity measured during MEG | 3 Hours
  as a result of altering cerebral perfusion in response to neurophysiologic stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Biyu He, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided